CLINICAL TRIAL: NCT04622865
Title: Randomized, Phase 2 Clinical Trial to Evaluate the Safety and Efficacy of Masitinib Combined With Isoquercetin, and Best Supportive Care in Hospitalized Patients With Moderate and Severe COVID-19
Brief Title: Masitinib Combined With Isoquercetin and Best Supportive Care in Hospitalized Patients With Moderate and Severe COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AB20001; 2020-001635-27 (EudraCT Number)
Record Dates: First submitted 2020-11-09; First posted 2020-11-10 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: SARS-CoV 2; COVID-19; Coronavirus Disease 2019
MeSH Terms: conditions — COVID-19 | interventions — masitinib; isoquercitrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Masitinib plus Isoquercetin plus Best Supportive Care (Experimental): Patients will receive oral masitinib dose of 3 mg/kg/day for 4 days then 4.5 mg/kg/day.
  The dose of isoquercetin will be 1 g/day by oral route. Best Supportive Care is best available therapy at the choice of the investigator, including, but not limited to, oxygenation, analgesics, anti-thrombotics, anti-viral drugs, or biologics drugs.
  Interventions: Drug: Masitinib; Drug: Isoquercetin; Drug: Best Supportive Care
- Best Supportive Care (Active Comparator): Best Supportive Care is best available therapy at the choice of the investigator, including, but not limited to, oxygenation, analgesics, anti-thrombotics, anti-viral drugs, or biologics drugs.
  Interventions: Drug: Best Supportive Care

INTERVENTIONS:
Drug: Masitinib — Masitinib is a small molecule drug that selectively inhibits specific tyrosine kinases such as colony-stimulating factor 1 receptor (CSF1R), c-Kit, LYN, FYN, and platelet-derived growth factor receptor (PDGFR) α and β, in the submicromolar range.
  Other Names: AB1010
  Arms: Masitinib plus Isoquercetin plus Best Supportive Care
Drug: Isoquercetin — Isoquercetin is a flavonoid, derivative of quercetin. Isoquercetin is rapidly hydrolyzed to quercetin.
  Other Names: quercetin-3-O-glucoside; isotrifoliin
  Arms: Masitinib plus Isoquercetin plus Best Supportive Care
Drug: Best Supportive Care — Best Supportive Care is best available therapy at the choice of the investigator, including, but not limited to, oxygenation, analgesics, anti-thrombotics, anti-viral drugs or biologics drugs.
  Other Names: BSC

SUMMARY:
Study objective is to evaluate the efficacy of the combination of masitinib and isoquercetin in adult hospitalized patients with moderate and severe COVID-19.

DETAILED DESCRIPTION:
COVID-19 is a respiratory disease caused by a novel coronavirus (SARS-CoV-2) that is associated with substantial morbidity and mortality. There is currently no vaccine to prevent COVID-19 or infection with SARS-CoV-2 or therapeutic agent to treat COVID-19.

Many patients with moderate and severe COVID-19, develop a "cytokine storm" that leads to severe pulmonary inflammation and various thrombotic events associated with acute respiratory distress syndrome (ARDS) and potentially death. The combination of masitinib and isoquercetin may prevent the development of these two complications. Masitinib is a potent blocker of mast cells and macrophages that are contributors to the cytokine storm. Isoquercetin inhibits disulfide isomerase (PDI), an enzyme directly involved in the formation of clots, and also decreases D-Dimer, a predictor of COVID-19 thrombosis severity.

The primary objective of this study is to evaluate efficacy of the masitinib and isoquercetin combination in moderate and severe COVID-19 patients. The primary endpoint is subject clinical status at day 15, using a 7-point ordinal scale that is defined as follows: 1. Not hospitalized, no limitations on activities; 2.Not hospitalized, limitation on activities; 3. Hospitalized, not requiring supplemental oxygen; 4. Hospitalized, requiring supplemental oxygen; 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices; 6. Hospitalized, on invasive mechanical ventilation or ECMO; 7. Death.

ELIGIBILITY:
Inclusion Criteria:

* Has laboratory-confirmed SARS-CoV-2 infection
* Hospitalized patients for the treatment of COVID pneumopathy
* Patients not requiring ICU at admission with moderate and severe pneumopathy according to the OMS Criteria of severity of COVID pneumopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Clinical status of patients at day-15 using a 7-point ordinal scale | 15 days
  Ordinal scale defined as follows: 1. Not hospitalized, no limitations on activities; 2.Not hospitalized, limitation on activities; 3. Hospitalized, not requiring supplemental oxygen; 4. Hospitalized, requiring supplemental oxygen; 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices; 6. Hospitalized, on invasive mechanical ventilation or ECMO; 7. Death.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Chanez, MD, Principal Investigator — Department of Respiratory Diseases, Aix-Marseille University, Marseille, France
Locations (6):
- France (6):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Le Tripode, Groupe hospitalier Pellegrin CHU de Bordeaux, Bordeaux
  - CHU Clermont-Ferrand: Site Gabriel-Montpied, Clermont-Ferrand
  - Hopital Nord, AP-HM, Marseille
  - CHR Orleans, Hopital de la Source, Orléans
  - Hopital Larrey, CHU du Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Durojaye OA, Okoro NO, Odiba AS, Nwanguma BC. MasitinibL shows promise as a drug-like analog of masitinib that elicits comparable SARS-Cov-2 3CLpro inhibition with low kinase preference. Sci Rep. 2023 Apr 28;13(1):6972. doi: 10.1038/s41598-023-33024-2. PMID 37117213
- [Derived] Latham BD, Oskin DS, Crouch RD, Vergne MJ, Jackson KD. Cytochromes P450 2C8 and 3A Catalyze the Metabolic Activation of the Tyrosine Kinase Inhibitor Masitinib. Chem Res Toxicol. 2022 Sep 19;35(9):1467-1481. doi: 10.1021/acs.chemrestox.2c00057. Epub 2022 Sep 1. PMID 36048877